CLINICAL TRIAL: NCT01478152
Title: A Single Center, Dose Finding, Safety, and Feasibility Study to Investigate the Effect of Ectoin® Inhalation Solution on Subjects With Mild Bronchial Asthma
Brief Title: Effect of Ectoin® Inhalation Solution on Subjects With Mild Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: K-AN
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma; Ectoin; Ectoine; FeNO; Metacholin; sRaw
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ectoin Inhalation Solution (Experimental): After baseline visit subjects will receive 0.9% saline inhalation solution for placebo. Patients will be instructed to inhale once daily with the AKITA2® APIXNEB® inhalation system for 5 - 7 days.
  The treatment phase with low dose of Ectoin® will follow subsequently without any washout phase. This treatment phase will be repeated for medium and a high Ectoin® dose. All doses of Ectoin® inhalation solution will be administered for 5 - 7 days without any washout phase. Sputum inductions will be conducted on the last but one day of placebo treatment phase and on the last but one day of treatment phase with the highest Ectoin® dose.
  Interventions: Other: Drug-like Medical Device: Ectoin Inhalation Solution

INTERVENTIONS:
Other: Drug-like Medical Device: Ectoin Inhalation Solution — After baseline visit subjects will receive 0.9% saline inhalation solution for placebo. Patients will be instructed to inhale once daily with the AKITA2® APIXNEB® inhalation system for 5 - 7 days.
  The treatment phase with low dose of Ectoin® will follow subsequently without any washout phase. This treatment phase will be repeated for medium and a high Ectoin® dose. All doses of Ectoin® inhalation solution will be administered for 5 - 7 days without any washout phase. To minimize circadian variations Methacholine challenge tests will be performed always at the approximately same time. Sputum inductions will be conducted on the last but one day of placebo treatment phase and on the last but one day of treatment phase with the highest Ectoin® dose.

SUMMARY:
In this single center, dose finding, safety study the effect of inhaled Ectoin® inhalation solution will be investigated in subjects with mild bronchial asthma. This dose-finding study will estimate the minimum effective dose and will assess the safe dosage, in terms of the quantity given to patients. The results will be compared to baseline measurements. The results regarding Sputum measurements will be compared to measurements after placebo administration.

DETAILED DESCRIPTION:
Based on the anti-inflammatory effects of inhaled Ectoin® shown in previous animal studies, this trial aims to investigate the effects in terms of a reduction of the unspecific bronchial hyperresponsiveness (BHR) to Methacholine challenge test on subjects with mild bronchial asthma. In addition, measurements of exhaled nitric oxide level as an indicator of bronchial inflammation will be investigated.

This study will focus primarily on safety and dose finding in 12 to 18 subjects with mild bronchial asthma.

After a screening visit, subjects will be treated with placebo, followed by increasing doses of Ectoin® (low, medium and high dose). All doses of Ectoin® inhalation solution and placebo will be administered for 5 - 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 - 65 years)
* FEV1 ≥ 80% of predicted for patient's normal value pre bronchodilator (according to European Coal and Steel Community reference values)
* Positive Methacholine challenge test (PD20 ≤ 0.5 mg)
* A general practitioner or consultant diagnosed mild bronchial asthma
* Non or ex smoker (for more than 6 months, pack years (PY) ≤ 5)

Exclusion Criteria:

* Pregnant or lactating females
* Participation in another clinical study in the previous month
* Severe concomitant disease which may have an impact on the study participation
* Hypersensibility against Ectoin®
* Patients who have had treatment with live attenuated vaccinations within 14 days prior to screening visit (Inactivated influenza vaccination is acceptable, provided it is not administered within 7 days prior to screening visit).
* Other respiratory diseases (e.g. Chronic obstructive pulmonary disease (COPD), cystic fibrosis, alpha-1-Antitrypsin deficiency, sarcoidosis, bronchiectasis, allergic alveolitis, tuberculosis, etc.)
* Upper and lower airway respiratory infection within 4 weeks prior to study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Dose of Metacholine needed to produce a 20% drop in FEV1 as reflection of airway hyperreagibility | 5 to 7 days
  Methacholine cumulative dose producing a 20% decrease in Forced Expiratory Volume in 1 second (FEV1) (defined as PD20)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, MD, Principal Investigator — Inamed Research GmbH
Locations (1):
- Inamed Research GmbH & Co KG, Gauting, Bavaria, Germany